CLINICAL TRIAL: NCT00434850
Title: Peritransplant Deoxyspergualin in Islet Transplantation in Type 1 Diabetes (CIT-03)
Brief Title: Peritransplant Deoxyspergualin in Islet Transplantation in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-03
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Insulin dependence; Hypoglycemia; Hyperglycemia unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — gusperimus; Antilymphocyte Serum; Daclizumab; Basiliximab; Sirolimus; Tacrolimus; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Pancreatic Islet Cells (Experimental): Participants in this study can receive up to three separate islet transplants. They will begin receiving antithymocyte globulin (ATG) and sirolimus 2 days prior to the first islet transplant. ATG will continue to be given until Day 2 post-transplant. Participants will continue taking sirolimus for the duration of the study. On the day of transplant, participants will receive DSG and etanercept, in addition to ATG and sirolimus. The DSG infusion will be administered over 3 hours and will immediately precede the islet transplant. Participants will continue receiving daily 3-hour infusions of DSG through Day 6 post-transplant. Etanercept will also be administered on Days 3, 7, and 10 post-transplant. Tacrolimus will be administered on Day 1 post-transplant and continued throughout the study.
  Interventions: Biological: Allogeneic Pancreatic Islet Cells; Drug: Deoxyspergualin; Biological: Antithymocyte globulin; Biological: Daclizumab or basiliximab; Drug: Sirolimus; Drug: Tacrolimus; Biological: Etanercept

INTERVENTIONS:
Biological: Allogeneic Pancreatic Islet Cells — Preparation of allogeneic pancreatic islet cells injected into the portal vein of the liver
Drug: Deoxyspergualin — An anti-inflammatory agent that blocks proinflammatory cytokine production and inhibits T-cells and B-cells and affects antigen presenting cells.
Biological: Antithymocyte globulin — Immunosuppressive that selectively depletes activated T-cells and depletes resting T-cells in a dose-dependent manner.
Biological: Daclizumab or basiliximab — Will replace antithymocyte globulin in all islet transplantations after the first one
Drug: Sirolimus — Maintenance immunosuppressive therapy
Drug: Tacrolimus — Maintenance immunosuppressive therapy
Biological: Etanercept — Blocks TNF-alpha which is toxic to islet cells

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to assess the safety and efficacy of deoxyspergualin (DSG), an immunosuppressant drug, on post-transplant islet function in people with type 1 diabetes who have not responded to intensive insulin therapy.

DETAILED DESCRIPTION:
Type 1 diabetes, also known as insulin-dependent diabetes, is a chronic disease in which the pancreas produces insufficient insulin to properly regulate blood sugar levels. Hypoglycemia, low blood sugar, and hyperglycemia, high blood sugar, can lead to significant complications in people with type 1 diabetes. Intensive insulin therapy has been shown to reduce the risk of chronic complications in people who achieve near normalization of glycemia. However, this therapy is labor intensive, difficult to implement, and associated with an increased frequency of severe hypoglycemia. Transplantation of islets from a healthy pancreas has been successful in restoring normal blood sugar levels and has led to initial insulin independence in people with type 1 diabetes. Rejection of these islets by the recipient's immune system, however, makes the treatment ineffective within a couple of years. Immunosuppressant drugs may be an effective way to maintain islet function post-transplant. The purpose of this study is to assess the safety and efficacy of an immunosuppressive regimen that includes DSG on post-transplant islet function in people with type 1 diabetes who have not responded to intensive insulin therapy. The study will also seek to improve the understanding of determinants of success and failure of islet transplants for type 1 diabetes.

Following screening procedures and 2 days prior to islet transplant, participants will be randomly assigned to either this Phase 2 trial or a multicenter Phase 3 trial. Participants in this study will receive up to three separate islet transplants. They will begin receiving antithymocyte globulin (ATG) and sirolimus 2 days prior to the first islet transplant. ATG will continue to be given until Day 2 post-transplant. Participants will continue taking sirolimus for the duration of the study. On the day of transplant, participants will receive DSG and etanercept, in addition to ATG and sirolimus. The DSG infusion will be administered over 3 hours and will immediately precede the islet transplant. Participants will continue receiving daily 3-hour infusions of DSG through Day 6 post-transplant. Etanercept will also be administered on Days 3, 7, and 10 post-transplant. Tacrolimus will be administered on Day 1 post-transplant and continued throughout the study.

Transplantations will involve an inpatient hospital stay and infusion of islets into a branch of the portal vein. Participants who do not achieve or maintain insulin independence by Day 75 post-transplant will be considered for a second islet transplant. Participants who remain dependent on insulin for longer than 1 month after the second transplant and who show partial graft function will be considered for a third transplant. Daclizumab or basiliximab will be used in place of ATG for the second and third transplants, if they are necessary. Participants who do not meet the criteria for a subsequent transplant and do not have a functioning graft will enter a reduced follow-up period.

There will be up to 21 study visits following each transplant. A physical exam, review of adverse events, blood collection, urine tests, and measures of immunosuppression levels will occur at most visits. An abdominal ultrasound and glomerular filtration rate testing will occur at some study visits. Participants will also self-test their glucose levels at least five times per day throughout the study. A 12-month follow-up period will take place after the participant's last transplant.

ELIGIBILITY:
Inclusion Criteria:

* Mentally stable and able to comply with study procedures
* Clinical history compatible with type 1 diabetes, with onset of disease at less than 40 years of age; insulin dependence for at least 5 years at study entry; AND sum of age and insulin-dependent diabetes duration of at least 28
* Absent stimulated C-peptide (less than 0.3 ng/ml) 60 and 90 minutes post mixed-meal tolerance test
* Involvement of intensive diabetes management, defined as:

  1. Self monitoring of glucose values no less than a mean of three times each day, averaged over each week
  2. Administration of three or more insulin injections each day or insulin pump therapy
  3. Under the direction of an endocrinologist, diabetologist, or diabetes specialist, with at least three clinical evaluations during the past 12 months prior to study enrollment
* At least one episode of severe hypoglycemia, defined as an event with one of the following symptoms: memory loss; confusion; uncontrollable behavior; irrational behavior; unusual difficulty in awakening; suspected seizure; seizure; loss of consciousness; or visual symptoms, in which the participant was unable to treat him/herself and which was associated with either a blood glucose level less than 54 mg/dl or prompt recovery after an oral carbohydrate, intravenous glucose, or glucagon administration in the 12 months prior to study enrollment.
* Reduced awareness of hypoglycemia. More information about this criterion, including the specific definition of hypoglycemia unawareness, is in the protocol.

Exclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m2 or weight less than or equal to 50 kg
* Insulin requirement of more than 1.0 IU/kg/day or less than 15 U/day
* HbA1c greater than 10%
* Untreated proliferative diabetic retinopathy
* Systolic blood pressure higher than 160 mmHg or diastolic blood pressure higher than 100 mmHg
* Measured glomerular filtration rate using iohexol of less than 80 ml/min/1.73m2. More information about this criterion is in the protocol.
* Presence or history of macroalbuminuria (greater than 300 mg/g creatinine)
* Presence or history of panel-reactive anti-HLA antibody levels greater than background by flow cytometry. More information about this criterion is in the protocol.
* Pregnant, breastfeeding, or unwilling to use effective contraception throughout the study and for 4 months after study completion
* Active infection, including hepatitis B virus, hepatitis C virus, HIV, or tuberculosis. More information about this criterion is in the protocol.
* Negative for Epstein-Barr virus by IgG determination
* Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection in the past year
* History of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known active alcohol or substance abuse
* Baseline Hgb below the lower limits of normal, lymphopenia, neutropenia, or thrombocytopenia
* History of Factor V deficiency
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy after transplantation or individuals with an INR greater than 1.5
* Severe coexisting cardiac disease, characterized by any one of the following conditions:

  1. Heart attack within the last 6 months
  2. Evidence of ischemia on functional heart exam within the year prior to study entry
  3. Left ventricular ejection fraction less than 30%
* Persistent elevation of liver function tests at the time of study entry
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with the ability to absorb oral medications
* Hyperlipidemia despite medical therapy, defined as fasting LDL cholesterol greater than 130 mg/dl (treated or untreated) and/or fasting triglycerides greater than 200 mg/dl
* Currently receiving treatment for a medical condition that requires chronic use of systemic steroids except for the use of less than or equal to 5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only
* Treatment with any anti-diabetic medication other than insulin within 4 weeks prior to study entry
* Use of any study medications within the past 4 weeks
* Received a live attenuated vaccine within the past 2 months
* Any medical condition that, in the opinion of the investigator, might interfere with safe participation in the trial
* Treatment with any immunosuppressive regimen at the time of enrollment.
* A previous islet transplant.
* A previous pancreas transplant, unless the graft failed within the first week due to thrombosis, followed by pancreatectomy and the transplant occurred more than 6 months prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2011-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Insulin-independent Subjects | 75 days following the first islet transplant

SECONDARY OUTCOMES:
Percent Reduction in Insulin Requirements | 75 days following the first and subsequent islet transplant
Hemoglobin A1c (HbA1c) | 75 days following the first and subsequent islet transplant
Mean Amplitude of Glycemic Excursions (MAGE) | 75 days following the first and subsequent islet transplant
Glycemic Lability Index (LI) | 75 days following the first and subsequent islet transplant
Ryan Hypoglycemia Severity Score (HYPO) | 75 days following the first and subsequent islet transplant
Basal (fasting) and 90-minute Glucose and C-peptide Results | 75 days following the first and subsequent islet transplant
  Derived from Mixed Meal Tolerance Test (MMTT)
Beta-score | 75 days following the first and subsequent islet transplant
  Assesses beta-cell function after islet transplantation
C-peptide: Glucose Creatinine Ratio | 75 days following the first and subsequent islet transplant
Acute Insulin Response to Glucose, Insulin Sensitivity, and Disposition Index | 75 days following the first and subsequent islet transplant
  Derived from the insulin-modified frequently sampled intravenous glucose tolerance (FSIGT) test
Glucose Variability and Hypoglycemia Duration | 75 days following the first and subsequent islet transplant
  Derived from the continuous glucose monitoring system (CGMS)
Quality of Life (QOL) Measure | 75 days following the first and subsequent islet transplant
Incidence of Worsening Retinopathy | 365 days following the first islet transplant
Proportion of Insulin-independent Subjects | 365 days following the first and final islet transplant
Percent Reduction in Insulin Requirements | 365 days following the first and final islet transplant
Hemoglobin A1c (HbA1c) | 365 days following the first and final islet transplant
Mean Amplitude of Glycemic Excursions (MAGE) | 365 days following the first and final islet transplant
Glycemic Lability Index (LI) | 365 days following the first and final islet transplant
Clarke Score | 365 days following the first and final islet transplant
  A hypoglycemia score
HYPO Score | 365 days following the first and final islet transplant
  A hypoglycemia score
Basal (fasting) and 90-minute Glucose and C-peptide | 365 days following the first and final islet transplant
  Derived from Mixed Meal Tolerance Test (MMTT)
Beta-score | 365 days following the first and final islet transplant
  Assesses beta-cell function after islet transplantation
C-peptide: Glucose Creatinine Ratio | 365 days following the first and final islet transplant
Quality of life (QOL) Measure | 365 days following the first and final islet transplant
Proportion of Subjects Receiving a Second Islet Cell Transplant | 365 days following the first islet transplant
Proportion of Subjects Receiving a Third Islet Cell Transplant | 365 days following the first and final islet transplant
Incidence and Severity of Adverse Events Related to the Islet Cell Transplant Procedure | 75 days and 365 days following the first and final islet cell infusion
Incidence and Severity of Adverse Events Related to the Immunosuppression Therapy | 75 days and 365 days following the first and final islet transplant
Incidence of a Change in the Immunosuppression Drug Regimen | 75 days and 365 days following the first and final islet cell transplant
Incidence of Immune Sensitization | 75 days and 365 days following the first and final islet transplant
  Defined by detecting anti-HLA antibodies not present prior to transplantation
Acute Insulin Response to Glucose, Insulin Sensitivity, and Disposition Index (DI) | 365 day following the first and final islet transplant
  Derived from the insulin-modified frequently sampled intravenous glucose tolerance (FSIGT) test

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Hering, MD, Principal Investigator — University of Minnesota; Xunrong Luo, MD, PhD, Principal Investigator — Northwestern University; Andrew Posselt, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of Californinia, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- See also: Click here for the Clinical Islet Transplantation Consortium Web site — http://www.CITIsletstudy.org